CLINICAL TRIAL: NCT04510948
Title: Patient Priority Care for Older Adults With Multiple Chronic Conditions Achieved Through Primary and Specialty Care Alignment
Brief Title: Patient Priority Care for Older Adults With Multiple Chronic Conditions
Acronym: PPC-CCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Yale University (Other); Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Ardeshir Hashmi, Center Director, Geriatrics, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-555
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Multiple Chronic Conditions
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: The aim of this project is to test, using a parallel group design involving 2 matched primary care sites, whether PPC decreases patient treatment burden and unwanted and unnecessary health care as well as assess what the value of this program is for patients.
Who Masked: Outcomes Assessor
Masking Description: Baseline and follow up interviews will be conducted by a rater blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Implementing Patient Priorities Care) (Experimental): Patient Priorities Care requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences (collectively referred to as health priorities). Participants will be contacted by a trained priorities facilitator in-person or over the phone to elicit their health priorities. This information will be documented in the PPC- GOALS AND PREFERENCES form in the EHR and shared with the clinicians who will then use the Patient Priorities Care approach with patients to inform and guide treatment decisions.
  Interventions: Behavioral: Patient Priorities Care
- Usual Care (Not implementing PPC) (No Intervention): Patients will receive routine clinical care.

INTERVENTIONS:
Behavioral: Patient Priorities Care — Patient Priorities Care (PPC) is an innovative approach to shared decision-making that draws from existing professional training.
  PPC requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences. This information will be collected and documented in the EHR by facilitators and shared with the clinicians who will then use the PPC approach with patients to inform and guide treatment decisions.
  The PCPs will be trained in decisional strategies that have been shown to help align care with patients' health priorities. While encouraged to use these decisional strategies, PCPs will be free to make the recommendations they feel most appropriate for each patient.
  This intervention has been developed to be integrated seamlessly into usual care.
  Other Names: PPC
  Arms: Intervention (Implementing Patient Priorities Care)

SUMMARY:
Healthcare for older adults with multiple chronic conditions (MCCs) is burdensome and of uncertain benefit, resulting in unwanted and unhelpful care. Patient Priorities Care (PPC) aligns care with patients' health priorities (i.e. the health outcomes most desired given the healthcare each is willing and able to receive). The aim of this project is to test, using a parallel group design involving 2 matched primary care sites, whether PPC decreases patient treatment burden and unwanted and unnecessary health care as well as assess what the value of this program is for patients.

DETAILED DESCRIPTION:
Healthcare for older adults with multiple chronic conditions (MCCs) is burdensome and of uncertain benefit, resulting in unwanted and unhelpful care. Patient Priorities Care (PPC) is an approach that aligns care with patients' health priorities (i.e. the health outcomes most desired given the healthcare each is willing and able to receive). PPC offers the opportunity to increase value by improving both outputs (desired health outcomes) and inputs (healthcare preferences) for these major users of healthcare.

We will employ a quasi-experimental, usual care (UC) group design, involving 2 primary care sites (1 PPC and 1 UC. Patients are assigned to intervention or usual care arms based on their primary care practice location. We will use analytic techniques (e.g., inverse propensity score weighting) designed to reduce selection bias and balance PPC and UC sites in terms of baseline characteristics. Data collection will occur through quantitative and qualitative interviews and health encounter information in the Electric Health Record(EHR).

Patient Priorities Care requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with goals and priorities to achieve patients' health outcome goals and reduce the burden of multi-morbidity. Participants will be enrolled in the Patient Priorities Care Program and speak with a trained health priorities facilitator to elicit their healthcare preferences and health outcome goals, which together constitute their health priorities. This information will be documented, entered into the EHR, and shared with the clinicians who will then use the Patient Priorities Care approach with patients to inform and guide treatment decisions. Patients will participate in the program and be followed for up to one year from the health priorities identification visit.

To determine the value of PPC, comparable primary care sites within the Cleveland Clinic will be assigned to PPC or Usual care (UC). Clinicians and staff at the PPC site will be trained to identify and align decision-making with the health priorities of older adults with MCCs. Value will be compared using patient and provider-reported outcomes, healthcare utilization, and possibly costs at PPC and UC sites.

The ultimate goal of our work is to implement and evaluate this approach to care for older adults with multiple chronic conditions that focuses on what matters most to them and is less fragmented and burdensome, resulting in better quality and outcomes at lower cost. This study will focus on evaluating practice change at test sites at the Cleveland Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Age 66 and older
2. In the Cleveland Clinic patient population
3. In the clinician practices selected as intervention or usual care practice sites
4. Clinically identified by: Those who meet any of several criteria i. 3 chronic conditions (See appendix 0 for the complete list) ii. 10 medications iii. >2 ED visits over the past year iv. >1 hospitalization (or >10 days in hospital) v. receive any care coordination services vi. 2 specialists over past year

Exclusion Criteria:

1. In hospice or meeting hospice criteria for any condition
2. Advanced dementia or moderate to profound intellectual disabilities
3. Not English speaking
4. Nursing home resident

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 264 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Hashmi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Lakewood Family Health Center, Lakewood, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Dedientified data may be shared on a case-by-case basis after compliance and regulatory approval have been obtained.
Time Frame: After publication. Data will be retained for a period of six year after study closure.
Access Criteria: Access will be provided on a case-by-case basis pending approval by the Cleveland Clinic IRB and law department.

REFERENCES:
- [Background] Boyd C, Smith CD, Masoudi FA, Blaum CS, Dodson JA, Green AR, Kelley A, Matlock D, Ouellet J, Rich MW, Schoenborn NL, Tinetti ME. Decision Making for Older Adults With Multiple Chronic Conditions: Executive Summary for the American Geriatrics Society Guiding Principles on the Care of Older Adults With Multimorbidity. J Am Geriatr Soc. 2019 Apr;67(4):665-673. doi: 10.1111/jgs.15809. Epub 2019 Mar 10. PMID 30663782
- [Background] Tinetti ME, Naik AD, Dindo L, Costello DM, Esterson J, Geda M, Rosen J, Hernandez-Bigos K, Smith CD, Ouellet GM, Kang G, Lee Y, Blaum C. Association of Patient Priorities-Aligned Decision-Making With Patient Outcomes and Ambulatory Health Care Burden Among Older Adults With Multiple Chronic Conditions: A Nonrandomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1688-1697. doi: 10.1001/jamainternmed.2019.4235. PMID 31589281
- [Background] Z. Zhao, "Using matching to estimate treatment effects: Data requirements, matching metrics, and Monte Carlo evidence," in Review of Economics and Statistics, 2004, doi: 10.1162/003465304323023705.
- [Background] D. B. Rubin, "Using Multivariate Matched Sampling and Regression Adjustment to Control Bias in Observational Studies," J. Am. Stat. Assoc., 1979, doi: 10.1080/01621459.1979.10482513.
- [Background] Tran VT, Harrington M, Montori VM, Barnes C, Wicks P, Ravaud P. Adaptation and validation of the Treatment Burden Questionnaire (TBQ) in English using an internet platform. BMC Med. 2014 Jul 2;12:109. doi: 10.1186/1741-7015-12-109. PMID 24989988
- [Background] Hahn EA, Kallen MA, Jensen RE, Potosky AL, Moinpour CM, Ramirez M, Cella D, Teresi JA. Measuring social function in diverse cancer populations: Evaluation of measurement equivalence of the Patient Reported Outcomes Measurement Information System(R) (PROMIS(R)) Ability to Participate in Social Roles and Activities short form. Psychol Test Assess Model. 2016 Jun 27;58(2):403-421. PMID 30221102
- [Background] Groff AC, Colla CH, Lee TH. Days Spent at Home - A Patient-Centered Goal and Outcome. N Engl J Med. 2016 Oct 27;375(17):1610-1612. doi: 10.1056/NEJMp1607206. No abstract available. PMID 27783911
- [Background] Russell LB, Ibuka Y, Carr D. How Much Time Do Patients Spend on Outpatient Visits?: The American Time Use Survey. Patient. 2008 Jul 1;1(3):211-22. doi: 10.2165/1312067-200801030-00008. PMID 22272927
- [Background] Forcino RC, Barr PJ, O'Malley AJ, Arend R, Castaldo MG, Ozanne EM, Percac-Lima S, Stults CD, Tai-Seale M, Thompson R, Elwyn G. Using CollaboRATE, a brief patient-reported measure of shared decision making: Results from three clinical settings in the United States. Health Expect. 2018 Feb;21(1):82-89. doi: 10.1111/hex.12588. Epub 2017 Jul 5. PMID 28678426
- [Background] Blaum CS, Rosen J, Naik AD, Smith CD, Dindo L, Vo L, Hernandez-Bigos K, Esterson J, Geda M, Ferris R, Costello D, Acampora D, Meehan T, Tinetti ME. Feasibility of Implementing Patient Priorities Care for Older Adults with Multiple Chronic Conditions. J Am Geriatr Soc. 2018 Oct;66(10):2009-2016. doi: 10.1111/jgs.15465. Epub 2018 Oct 3. PMID 30281777
- [Background] Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Stat Med. 2015 Dec 10;34(28):3661-79. doi: 10.1002/sim.6607. Epub 2015 Aug 3. PMID 26238958
- [Background] D. B. Rubin, "Using propensity scores to help design observational studies: Application to the tobacco litigation," Matched Sampl. Causal Eff., pp. 365-382, 2006, doi:
- [Background] Stuart EA. Matching methods for causal inference: A review and a look forward. Stat Sci. 2010 Feb 1;25(1):1-21. doi: 10.1214/09-STS313. PMID 20871802
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] D. Rubin, Multiple Imputation for Nonresponse in Surveys. Wiley, 1987.
- [Background] J. Cohen, Statistical Power Analysis for the Behavioral Sciences. Hillsdale, New Jersey, 1988.
- [Background] Tinetti M, Dindo L, Smith CD, Blaum C, Costello D, Ouellet G, Rosen J, Hernandez-Bigos K, Geda M, Naik A. Challenges and strategies in patients' health priorities-aligned decision-making for older adults with multiple chronic conditions. PLoS One. 2019 Jun 10;14(6):e0218249. doi: 10.1371/journal.pone.0218249. eCollection 2019. PMID 31181117
- [Derived] Tinetti ME, Hashmi A, Ng H, Doyle M, Goto T, Esterson J, Naik AD, Dindo L, Li F. Patient Priorities-Aligned Care for Older Adults With Multiple Conditions: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352666. doi: 10.1001/jamanetworkopen.2023.52666. PMID 38261319
- See also: Patient Priorities Care helps patients and clinicians focus all decision-making and healthcare on what matters most: patients' own health priorities. It was developed by clinicians, patients, caregivers, health system leaders, and payers. — https://patientprioritiescare.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between August 14, 2020 - May 14, 2021. The study followed a nonrandomized controlled trial design. One primary care site within Cleveland Clinic's multisite Primary Care Practice was selected as the PPC site. The UC site was identified as the optimal match to the PPC site using a multivariate matching procedure which calculated the multivariate distance between the PPC site and 11 potential UC sites.
Units Other Than Participants: Clinic
Period: Overall Study
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
Started | 129; 1 Clinic | 135; 1 Clinic
Completed | 116; 1 Clinic | 113; 1 Clinic
Not Completed | 13; 0 Clinic | 22; 0 Clinic

BASELINE CHARACTERISTICS:
Population: The number above includes respondents with some missing data. Although not all respondents answered all questions, all participants who responded completely at least one scale are included here. Raw numbers are reported.
Groups:
- Intervention (Implementing Patient Priorities Care): Patient Priorities Care (PPC) requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences (collectively referred to as health priorities). Participants will be contacted by a trained priorities facilitator in-person or over the phone to elicit their health priorities. This information will be documented in the PPC-GOALS AND PREFERENCES form in the EHR and shared with the clinicians who will then use the Patient Priorities Care approach with patients to inform and guide treatment decisions.
  PPC is an innovative approach to shared decision-making that draws from existing professional training.
  PPC requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences. This information will be collected and documented in the EHR by facilitators and shared with the clinicians who will then use the PPC approach with patients to inform and guide treatment decisions.
  The PCPs will be trained in decisional strategies that have been shown to help align care with patients' health priorities. While encouraged to use these decisional strategies, PCPs will be free to make the recommendations they feel most appropriate for each patient.
  This intervention has been developed to be integrated seamlessly into usual care.
- Usual Care (Not Implementing PPC): Patients will receive routine clinical care. No study intervention was provided before or during their scheduled visit.
- Total: Total of all reporting groups
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC) | Total
Number analyzed (Participants) | 129 | 135 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated based on DOB documented in the EHR, and at the time of baseline visit date. Population: Total is not 264 because of missing data.
  years
    number analyzed (Participants) | 125 | 134 | 259
    (all) | 75.5 (6.4) | 75.4 (6.1) | 75.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — the count is based on legal sex documented in the EHR. Population: there were missing data in the outcomes.
  Participants
    number analyzed (Participants) | 127 | 135 | 262
    Female | 54 | 66 | 120
    Male | 73 | 69 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants] — Results are based on EHR documents but variable was updated when different race was reported during phone interview. Population: One participant did not answer.
  Participants
    number analyzed (Participants) | 128 | 135 | 263
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 1 | 11
    White | 110 | 129 | 239
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 5 | 3 | 8
Education high school or less [Count of Participants; unit: Participants] — Based on self-reported education level during the phone interview. Population: Not all respondents answered all questions. Raw numbers are reported.
  Participants
    number analyzed (Participants) | 124 | 132 | 256
    (all) | 25 | 46 | 71
Medicare Advantage [Count of Participants; unit: Participants] — Based on EHR data (Financial class). Population: Not all respondents answered all questions. Raw numbers are reported.
  Participants
    number analyzed (Participants) | 126 | 135 | 261
    (all) | 59 | 63 | 122
Lives alone [Count of Participants; unit: Participants] — Based on self-report during phone interview. Population: Not all respondents answered all questions. Raw numbers are reported.
  Participants
    number analyzed (Participants) | 125 | 132 | 257
    (all) | 54 | 40 | 94
5-Word recall score [Mean (Standard Deviation); unit: words] — Adapted version of MoCA memory recall section was used during the baseline interview. Scores are based on number of words correctly recalled by participants after completing TBQ and PROMIS scales, typically, 5-10 minutes between.
  Total is not 264 because of missing data. Some patients declined to perform the task. Population: Score ranges between 0 to 5. Higher score represents better cognition. Some participants declined to perform this task.
  words
    number analyzed (Participants) | 118 | 131 | 249
    (all) | 3.4 (1.4) | 3.7 (1.4) | 3.6 (1.4)
PROMIS physical health [Mean (Standard Deviation); unit: units on a scale] — PROMIS Scale v1.2 - Global Health raw score is reported here. Physical health score was calculated by summing the responses for Global03, Global06, Global07r, and Global08r. This subscale raw score ranges from 4 to 20, the higher score represents better state of physical health.
  Total is not 264 because of missing data. Only patients who responded all items are included here. Population: Not all respondents answered all questions. Raw numbers are reported.
  units on a scale
    number analyzed (Participants) | 119 | 131 | 250
    (all) | 14.8 (2.9) | 14.3 (2.7) | 14.6 (2.8)
PROMIS mental health [Mean (Standard Deviation); unit: units on a scale] — PROMIS Scale v1.2 - Global Health raw score is reported here. Mental health score was calculated by summing the responses for Global 02, Global04, Global05, and Global10r. This subscale raw score ranges from 4 to 20, the higher score represents better state of mental health.
  Total is not 264 because of missing data. Only patients who responded all items are included here. Population: Not all respondents answered all questions. Raw numbers are reported.
  units on a scale
    number analyzed (Participants) | 119 | 131 | 250
    (all) | 14.3 (2.9) | 13.9 (2.8) | 14.1 (2.8)
The Treatment Burden Questionnaire (TBQ) score [Mean (Standard Deviation); unit: units on a scale] — The Treatment Burden Questionnaire (TBQ) aims to assess treatment burden in different condition and treatment contexts. The TBQ score ranges between 0 and 130, indicating the level of treatment burden a patient experiences. Higher scores indicate a higher level of burden. Population: Not all respondents answered all questions. Raw numbers are reported.
  units on a scale
    number analyzed (Participants) | 121 | 128 | 249
    (all) | 12.2 (12.6) | 10.3 (10.7) | 11.2 (11.7)
CollaboRATE top score [Count of Participants; unit: Participants] — higher score denoting greater perceived shared decision-making; dichotomized as 100 vs <100, with 100 being the percentage of participants who reported the top score of all 3 items. Population: Not all respondents answered all questions. Raw numbers are reported.
  Participants
    number analyzed (Participants) | 111 | 127 | 238
    (all) | 48 | 60 | 108
Number of chronic conditions, mean (+/- SD) [Mean (Standard Deviation); unit: condition(s)] — Count of 18 chronic conditions (based on Centers for Medicare and Medicaid Services' Chronic Conditions Warehouse International Statistical Classification of Diseases and Related Health Problems, Tenth Revision algorithms) were ascertained from the EHR. Population: The number reported here is based on EHR data.
  condition(s) | 6.0 (2.3) | 6.1 (2.1) | 6.1 (2.2)
Heart failure [Count of Participants; unit: Participants] — presence of heart failure Population: The number reported here is based on EHR data.
  Participants | 17 | 19 | 36
COPD [Count of Participants; unit: Participants] — presence of chronic lung disease Population: The number reported here is based on EHR data.
  Participants | 36 | 29 | 65
Number or oral prescription medications for chronic conditions, mean (+/- SD) [Mean (Standard Deviation); unit: medication(s)] — number of prescribed medication were ascertained from the EHR. Population: The number reported here is based on EHR data.
  medication(s) | 8.5 (3.9) | 8.0 (3.0) | 8.2 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Burden
Description: Change in patient score on 'Treatment Burden Questionnaire' (TBQ, score range 0-150, Cronbach's alpha=0.90) Lower score reflects less perceived treatment burden.
Time Frame: from baseline to follow-up at 8-9 months
Population: The baseline outcome is included to illustrate weighted balance of covariate before PPC is introduced, and the P values for the baseline outcome comparison are based on weighted and imputed data (same as the adjusted P values in Table 1).Of note, the baseline value of the outcome was included in outcome models at follow-up. Therefore, the difference between estimates for baseline and follow-up is not necessarily equal to the effect size reported.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Intervention (Implementing Patient Priorities Care): Patient Priorities Care requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences (collectively referred to as health priorities). Participants will be contacted by a trained priorities facilitator in-person or over the phone to elicit their health priorities. This information will be documented in the PPC-GOALS AND PREFERENCES form in the EHR and shared with the clinicians who will then use the Patient Priorities Care approach with patients to inform and guide treatment decisions.
  Patient Priorities Care: Patient Priorities Care (PPC) is an innovative approach to shared decision-making that draws from existing professional training.
  PPC requires the elicitation and documentation of patient health outcome goals and care preferences and the alignment of clinical care with health goals and healthcare preferences. This information will be collected and documented in the EHR by facilitators and shared with the clinicians who will then use the PPC approach with patients to inform and guide treatment decisions.
  The PCPs will be trained in decisional strategies that have been shown to help align care with patients' health priorities. While encouraged to use these decisional strategies, PCPs will be free to make the recommendations they feel most appropriate for each patient.
  This intervention has been developed to be integrated seamlessly into usual care.
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
Number analyzed (Participants) | 109 | 111
score on a scale
  Baseline | 11.9 [10.3 to 13.6] | 11.6 [9.3 to 14.0]
  Follow up | 12.7 [10.0 to 15.5] | 17.9 [13.1 to 22.7]

2. Primary Outcome: Achievement of Desired Activities
Description: Patient score on PROMIS Ability to Participate in Social Roles and Activities Shot Form 6a (score range 6-30; Cronbach's alpha = 0.98) Higher score reflects more social participation.
Time Frame: at follow-up (8-9 months) The scale instructions do not reference timeframe.
Population: PROM IS Social Roles and Activities was inadvertently left out of the baseline interview.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
Number analyzed (Participants) | 97 | 88
score on a scale | 21.9 [20.6 to 23.1] | 21.6 [20.2 to 22.9]

3. Primary Outcome: Health Care Utilization Defined by Healthcare Contact Days
Description: Number of health care contact days defined as number of ED visits, days in hospital +.5*number of outpatient encounters for procedures, tests, healthcare visits.
Time Frame: from 3 months prior to 12 months following baseline interview
Population: Baseline refers to 90 days before enrollment; follow-up refers to 365 days after enrollment. Baseline measures of nonhealthy days include only encounter days.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
Number analyzed (Participants) | 129 | 135
days
  Baseline | 0.7 [0.4 to 1.0] | 0.7 [0.4 to 1.0]
  Follow up | 8.7 [3.8 to 13.7] | 13.4 [6.6 to 20.1]

4. Secondary Outcome: Shared Decision Making and Goal Ascertainment
Description: Change in patient score on CollaboRATE tool (score 0-100, Cronbach's alpha=0.89) from baseline to follow-up up at 8-9 months and response to Cleveland Clinic ACO survey item "When starting a new medication, did your provider ask what you thought was best for you?" Scores are dichotomized 100 vs. <100 with 100 being the percent of participants who reported the top score of all three items.
Time Frame: at 8-9 months follow-up
Population: All results reflect doubly robust imputed models. Variables used in propensity weighting included race, gender, education, and baseline measures of age, living alone, insurance, cognitive status, number of oral prescription medications, number of chronic conditions, heart failure, COPD, baseline PROMIS mental health and physical health, baseline TBQ, baseline CollaboRATE, baseline ACO shared prescribing decision-making quality measure, and Nonhealthy Days in 90 days prior to enrollment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
Number analyzed (Participants) | 129 | 135
score on a scale
  Baseline | 46.3 [36.5 to 56.5] | 47.7 [37.9 to 57.8]
  Follow up | 58.5 [45.6 to 70.3] | 61.9 [50.9 to 71.8]

ADVERSE EVENTS:
Time Frame: From baseline and up to 1 year from baseline
Description: This is a minimal risk study using data collected for routine clinical practice and survey research.
Arm/Group | Intervention (Implementing Patient Priorities Care) | Usual Care (Not Implementing PPC)
All-Cause Mortality (participants affected / at risk) | 3/129 | 5/135
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/135
Other Adverse Events (participants affected / at risk) | 0/129 | 0/135

LIMITATIONS AND CAVEATS:
1) Despite careful site selection by propensity-adjusted analyses, potential unmeasured confounders and persistent recruitment disparities despite efforts. 2) Methodological constraints and the impact of the COVID-19 pandemic (delays, disruptions, and reduced sample size) further limit generalizability and statistical power. 3) Participant enrollment issues and 9-month follow-up limitations add complexities. 4) While promising, the study's long-term impact on health outcomes remains uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT04510948/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04510948/SAP_001.pdf
  • Informed Consent Form (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT04510948/ICF_002.pdf